CLINICAL TRIAL: NCT07199543
Title: Palatability Study of Five Formulations of Benzydamine HCl Lozenges
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 030(F/b)MD21257
Record Dates: First submitted 2025-09-09; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers; Palatability; To Test the Palatability of a New Flavour and Four Commercially Available Flavours
Keywords: Palatability test
MeSH Terms: interventions — Benzydamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Healthy adult (Experimental): A single oral dose (one lozenge) of each investigational medicinal product was administered to healthy adult in two study periods
  Interventions: Drug: benzydamine HCl
- Group 2: Paediatric volunteers (Experimental): A single oral dose (one lozenge) of each investigational medicinal product was administered to paediatric volunteers in two study periods
  Interventions: Drug: benzydamine HCl

INTERVENTIONS:
Drug: benzydamine HCl — The investigational medicinal products were tasted during two study ambulatory visits, separated by a wash-out of at least 3 days

SUMMARY:
This is a palatability study on 60 healthy adult and 60 healthy children with 5 different aroma of Lozenges. They will keep the lozenge in their mouth (without swallowing, chewing or breaking) for 10 seconds and then they will eject it. Palatability will be evaluated by the study participants 15 min after each investigational medicinal product ejection using a questionnaire. It will include common terms used to describe the formulation's taste, aftertaste and texture, and a hedonic 7-point facial scale used to quantitate the sensory experiences (i.e., pleasantness of the formulation taste, smell, aftertaste, texture and overall evaluation). A numeric score will be assigned for each provided reply.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, adults must fulfil all these criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Gender, age: any gender, 18-55 years old inclusive
3. Body Mass Index: 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-99 bpm, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
6. Contraception and fertility (females only): females of child-bearing potential must be using at least one of the following reliable methods of contraception:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
   2. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner
   5. True abstinence Periodic abstinence, lactational, amenorrhea, and withdrawal are not acceptable.

Females of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted.

For all females, pregnancy test result must be negative at screening and at visit 3.

To be enrolled in this study, minors must fulfil all these criteria:

1. Informed consent and assent: signed written informed consent by at least one parent/legal representative.

   Signed written informed assent for 14-17 years old inclusive adolescents or written informed assent for 11-13 years old inclusive children or oral informed assent for 6-10 years old inclusive children
2. Gender, age: any gender, 6-17 years old inclusive
3. Body Mass Index: not classified as overweight based on the applicable body mass index chart for sex and age
4. Vital signs: systolic blood pressure, diastolic blood pressure and heart rate within the normal ranges suitable for age measured after 5 min at rest in the sitting position
5. Full comprehension: ability of the paediatric volunteer and parent/legal representative to comprehend the full nature and purpose of the study, including possible risks and side effects; ability of the paediatric volunteer and parent/legal representative to co-operate with the Investigator and to comply with the requirements of the entire study
6. Contraception and fertility (females of child-bearing potential only): females of child-bearing potential must be using at least one of the following reliable methods of contraception:

   1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
   2. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner
   5. True abstinence Periodic abstinenc, lactational, amenorrhea, and withdrawal are not acceptable. For all females of child-bearing potential, pregnancy test result must be negative at screening and at visit 3.

Exclusion Criteria:

* Adults and minors meeting any of these criteria will not be enrolled in the study:

  1. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
  2. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; ascertained or presumptive hypersensitivity to acetylsalicylic acid or other non-steroidal anti-inflammatory drugs; intolerance to some sugars; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the study participants safety
  3. Diseases: history of significant renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study, in particular phenylketonuria or asthma or both; nasopharyngitis, rhinitis, cold, dysosmia, dysgeusia, mouth lesions or any other oral mucosa alteration that may interfere with the aim of the study according to the Investigator's opinion
  4. Medications: medications, including over the counter medications and herbal remedies for 2 weeks before the start of the study that may interfere with the aim of the study according to the Investigator's opinion. Hormonal contraceptives for child-bearing potential females will be allowed
  5. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
  6. Diet: abnormal diets or substantial changes in eating habits in the 4 weeks before this study that may interfere with the aim of the study according to the Investigator's opinion.

     Adults meeting any of these exclusion/withdrawal criteria:
  7. Drug, alcohol, caffeine, tobacco: history of (within the past 12 months) or current drug, alcohol, caffeine or tobacco abuse
  8. Positive result at the urine drug test at screening or at visit 3
  9. Positive alcohol saliva test at screening or at visit 3
  10. Pregnancy (females only): positive or missing pregnancy test at screening or at visit 3, pregnant or breastfeeding females.

Adolescents/children (12-17 years old inclusive) meeting any of these exclusion/withdrawal criteria:

Drug, alcohol, caffeine, tobacco: history of or current drug or alcohol consumption and history of or current tobacco use, history of or current caffeine consumption 8. Drug test: positive result at the urine drug test at screening or at visit 3 9. Alcohol test: positive alcohol saliva test at screening or at visit 3 10. Pregnancy (females only): for post-menarche females, positive or missing pregnancy test at screening or at visit 3, pregnant or breast-feeding females.

Children (6-11 years old inclusive) meeting any of these exclusion/withdrawal criteria:

7. Drug, alcohol, caffeine, tobacco: history of or current drug, alcohol or coffee consumption or tobacco use 8. Pregnancy (females only): for post-menarche females, positive or missing pregnancy test at screening or at visit 3, pregnant or breast-feeding females.

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2025-04-13 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Palatability of a new flavour | 15 min after the investigational medicinal product ejection
  The palatability of a new flavour and four commercially available flavours of Benzydamine HCl 3 mg lozenges, tasted by healthy adult and paediatric volunteers will be evaluated by the study participants 15 min after each investigational medicinal product ejection using a questionnaire. It will include common terms used to describe the formulation's taste, aftertaste and texture, and a hedonic 7-point facial scale -Chen scale- in which descriptive replies are associated to images showing different facial expressions to allow the children to easily quantitate their sensory experiences (i.e., pleasantness of the formulation taste, smell, aftertaste, texture and overall evaluation).
  For the Chen scale, a numeric score will be assigned by the Investigator to each provided reply, as follows: Very bad = 1, Bad = 2, Just a little bad = 3, Not sure = 4, Just a little good = 5, Good = 6, Very good = 7.
  Palatability evaluation scores will be listed and summarised using tables of frequency.

SECONDARY OUTCOMES:
Safety data after administration | Minimum study duration for each subject will be 4 days, screening visit included
  Subjects' blood pressure and heart rate will be measured by the Investigator or his/her deputy after 5 min at rest (in sitting position) at screening and final visit/ETV. For adults, normality parameters are clearly defined in the inclusion criteria. For minors, the Investigator or his/her deputy will verify that the measured parameters will be within the normal ranges suitable for age.
Safety data after administration | Minimum study duration for each subject will be 4 days, screening visit included
  Physical examination: The physical examination will include subject's oral cavity inspection. Information about the physical examination will be recorded by the Investigator. Any abnormalities will be recorded. Significant findings/illnesses, reported after the start of the study and that meet the definition of an AE, will be recorded in the subject source documents.
  Date of the physical examination, overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) will be reported in the eCRF.
Safety data after administration | Minimum study duration for each subject will be 4 days, screening visit included
  Body weight and height: Body weight and height will be recorded at screening visit only. Subjects will be weighed (kg) lightly clothed without shoes. For adults, BMI will be calculated as weight [kg]/(height [m] x height [m]). For minors, BMI will be evaluated on the basis of the applicable body mass index chart for sex and age
Tolerability data after administration | Minimum study duration for each subject will be 4 days, screening visit included
  Subjects' blood pressure and heart rate will be measured by the Investigator or his/her deputy after 5 min at rest (in sitting position) at screening and final visit/ETV. For adults, normality parameters are clearly defined in the inclusion criteria. For minors, the Investigator or his/her deputy will verify that the measured parameters will be within the normal ranges suitable for age.
Tolerability data after administration | Minimum study duration for each subject will be 4 days, screening visit included
  Physical examination: The physical examination will include subject's oral cavity inspection. Information about the physical examination will be recorded by the Investigator. Any abnormalities will be recorded. Significant findings/illnesses, reported after the start of the study and that meet the definition of an AE, will be recorded in the subject source documents.
  Date of the physical examination, overall Investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant) and clinically significant abnormalities (if any) will be reported in the eCRF.
Tolerability data after administration | Minimum study duration for each subject will be 4 days, screening visit included
  Body weight and height: Body weight and height will be recorded at screening visit only. Subjects will be weighed (kg) lightly clothed without shoes. For adults, BMI will be calculated as weight [kg]/(height [m] x height [m]). For minors, BMI will be evaluated on the basis of the applicable body mass index chart for sex and age

CONTACTS AND LOCATIONS:
Locations (1):
- CROSS Research S.A. - Phase I Unit, Arzo, Switzerland, Switzerland